CLINICAL TRIAL: NCT05589675
Title: Evaluation of the Home Delivery of the Screening Kit, and Impact of a Prior Notification Among New Participants to the National Organized Colorectal Cancer Screening Program (Among New Participants Only)
Brief Title: Evaluation of a New Invitation Procedure to the French Organized Colorectal Cancer Screening Program
Acronym: KITCOLO22
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Responsible Party: Principal Investigator, Catherine Sauvaget, Dr, International Agency for Research on Cancer
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IEC/22-29
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; screening program; pilot project; randomised control trial; France
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a three-arm study with a parallel study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention arm (Experimental): Invitation letter to the screening program with the FIT test
  Interventions: Other: Dispatch of the screening test along the invitation letter to the national colorectal cancer screening program
- Intervention arm - sub study (Experimental): Prior notification to the new entrants, followed by an invitation letter to the screening program with the FIT test
  Interventions: Other: Dispatch of the screening test along the invitation letter to the national colorectal cancer screening program; Other: Sending of a prior notification to the new entrants of the national program
- Control arm (No Intervention): Invitation letter to visit its own GP who will deliver the FIT test

INTERVENTIONS:
Other: Dispatch of the screening test along the invitation letter to the national colorectal cancer screening program — The individuals eligible for the colorectal cancer screening program will receive at home an invitation letter to participate to the program along with a FIT test. The follow-up will be similar to the standard of care, i.e. reminder letters at 5 and 10 months if there is no participation, and reminders if no coloscopy after a positive FIT test
  Arms: Intervention arm; Intervention arm - sub study
Other: Sending of a prior notification to the new entrants of the national program — Dispatch of a notification, one month prior the dispatch of the screening test along the invitation letter. This intervention is among the new entrants to the national program
  Arms: Intervention arm - sub study

SUMMARY:
This is a randomized controlled trial comparing the effect on participation rates to colorectal cancer screening between an intervention arm (invitation letter to the screening program including a FIT test with or without prior notification) and a control arm with the standard of care (invitation letter to visit the GP who will deliver the FIT test).

DETAILED DESCRIPTION:
The participation to the national screening program for colorectal cancer in France is low. In order to improve the performances of its organized program, the National Cancer Institute is planning to modify the invitation procedure. This is a pilot project and if an improvement in the program performances is reported, the invitation procedure may be scaled up.

Eligible individuals for colorectal cancer screening will be identified by the Regional Cancer Screening Coordinating Centre and randomized into the intervention or control arms. They will be followed for FIT test submission to the central laboratory (participation to screening). Those who did not send their test will receive reminder letters. Those who had a positive FIT test will be followed up for coloscopy referral, and result of the coloscopy. Comparison of the participation rates to screening program and to coloscopy among those with a positive FIT test will be compared between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 50 to 74 years old
* Living in the study area (Departments of Ardennes, Meurthe-et-Moselle, and Moselle, France)
* At moderate risk of colorectal cancer, i.e. eligible to the organised programme and receiving the first invitation of the screening round (not a reminder letter)

Exclusion Criteria:

* Outside the target age (less than 50 years old, or 75 years and more)
* Receiving the reminder letter
* At high or very high risk of colorectal cancer

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64500 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Participation rates to the screening program | 2 years
  Comparison of the participation rate to the screening program between the intervention and the control arms

SECONDARY OUTCOMES:
Referral rates to coloscopy among those FIT positive | 2 years
  Comparison of the referral rates to coloscopy between the intervention and the control arms
Participation rates to the screening program | 2 years
  Comparison of the participation rates to the screening program between the individuals aged 50-52 of the Intervention1 and the Intervention sub-study arms

CONTACTS AND LOCATIONS:
Overall Officials: Maurice TANGUY, MD, Principal Investigator — Regional Cancer Screening Coordinating Centre, Meurthe-et-Moselle site, Nancy, France; Myriam GUERBAZ SOMMI, MD, Principal Investigator — Regional Cancer Screening Coordinating Centre, Moselle site, Metz, France; Jean BOTO KEKY, MD, Principal Investigator — Regional Cancer Screening Coordinating Centre, Ardennes site, Charleville-Mézières, France
Locations (3):
- France (3):
  - Regional Cancer Screening Coordinating Centre, Ardennes site, Charleville-Mézières, Ardennes
  - Regional Cancer Screening Coordinating Centre, Meurthe-et-Moselle Site, Nancy, Meurthe-et-Moselle
  - Regional Cancer Screening Coordinating Centre, Moselle Site, Metz, Moselle

IPD SHARING:
Plan to Share IPD: No